CLINICAL TRIAL: NCT05174052
Title: Dapagliflozin in Patients With Atrial Fibrillation
Brief Title: Dapagliflozin in Patients With Atrial Fibrillation (DAPA-AF)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13694
Record Dates: First submitted 2021-10-21; First posted 2021-12-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Diabetes Mellitus; Atrial Fibrillation
MeSH Terms: conditions — Diabetes Mellitus; Atrial Fibrillation | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: This is a randomized, double blind, placebo-controlled trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control Arm (Placebo) (Placebo Comparator): Subjects will take 1 blinded tablet of placebo drug dosed once daily, per the randomization scheme.
  Interventions: Drug: Placebo
- Intervention Arm (Dapagliflozin) (Active Comparator): A block randomization method will be use to randomize subjects to treatment with dapagliflozin 10 mg once daily. Subjects will take 1 blinded tablet of study drug (dapagliflozin) dosed once daily, per the randomization scheme
  Interventions: Drug: Dapagliflozin 10Mg Tab

INTERVENTIONS:
Drug: Dapagliflozin 10Mg Tab — Subjects will take 1 blinded tablet of study drug (dapagliflozin 10 mg) dosed once daily.
  Arms: Intervention Arm (Dapagliflozin)
Drug: Placebo — Subjects will take 1 blinded capsule of placebo drug dosed once daily
  Arms: Control Arm (Placebo)

SUMMARY:
The study will investigate the effect of Dapagliflozin on atrial fibrillation (AF) burden. AF burden will be defined as the percent of time spent in AF over a 2-week period, assessed by noninvasive continuous heart rhythm monitoring at baseline and at 3 months, quality of life (QOL) and validated echocardiographic indices of atrial myopathy. This knowledge will enable us to study the therapeutic potential of SGLT2i as a novel adjunct treatment for patients with DM and AF. Patients with paroxysmal AF (AF that terminates spontaneously or with intervention within seven days of onset) and DM and randomize them to Dapagliflozin or placebo. Continuous heart rhythm monitoring patch for AF burden will be used, measure of QOL with the help of AF Effect on Quality-of-life survey and perform an echocardiogram with measurement of left atrial volume index, left atrial strain and atrial tissue dopplers. All measurements will be performed at baseline and at study completion. The central hypothesis is that SGLT2i will lead to reduced AF burden that will translate into improvement in QOL, and the underlying mechanism is improvement in atrial myopathy.

DETAILED DESCRIPTION:
Patients with diabetes mellitus (DM) and atrial fibrillation (AF) represent a high-risk cohort that is at an increased risk of cardiovascular complications as compared to AF patients without DM. Sodium-glucose cotransporter 2 inhibitors (SGLT2i) are a new class of diabetic drugs and large clinical trials have established their multiple cardiovascular benefits. However, none of these clinical trials studied AF as a primary outcome. SGLT2i have multiple properties that can be protective against AF and the role of SGLT2i in preventing recurrent AF remains an important knowledge gap.

In this translational research proposal, we aim to fill this knowledge gap by studying the effect of Dapagliflozin on AF burden. AF burden will be defined as the percent of time spent in AF over a 2-week period, assessed by noninvasive continuous heart rhythm monitoring at baseline and at 3 months, quality of life (QOL) and validated echocardiographic indices of atrial myopathy. This knowledge will enable us to study the therapeutic potential of SGLT2i as a novel adjunct treatment for patients with DM and AF. Patients with paroxysmal AF (AF that terminates spontaneously or with intervention within seven days of onset) and DM will be enrolled. Subjects will be randomized to Dapagliflozin or placebo. Continuous heart rhythm monitoring patch for AF burden, measure QOL with the help of AF Effect on Quality-of-life survey and perform an echocardiogram with measurement of left atrial volume index, left atrial strain and atrial tissue dopplers. All measurements will be performed at baseline and at study completion. Our central hypothesis is that SGLT2i will lead to reduced AF burden that will translate into improvement in QOL, and the underlying mechanism is improvement in atrial myopathy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with DM
* Paroxysmal AF

Exclusion Criteria:

* Type 1 DM,
* Symptoms of hypotension or systolic blood pressure <90mmHg,
* Severe renal impairment with eGFR<30mL/minute/1.73m2,
* History of lower limb amputation,
* Hypersensitivity to Dapagliflozin,
* Currently taking any SGLT2i,
* Pregnancy,
* Currently taking anti-arrhythmic drugs
* Undergoing catheter ablation will be excluded

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
The effect of Dapagliflozin on change in burden of atrial fibrillation | Baseline and 3 months
  To determine the effect of Dapagliflozin on change in AF burden in patients with AF and DM. AF burden will be defined as the percent of time spent in AF over a 2-week period, assessed by noninvasive continuous heart rhythm monitoring at baseline and at 3 months. The AF burden between Dapagliflozin vs Placebo will be compared.

SECONDARY OUTCOMES:
Effect of Dapagliflozin on change in AF Effect on Quality of Life Survey | Baseline and 3 months
  To determine the effect of Dapagliflozin on change in quality of life in patients with AF and DM. AF Effect on Quality of Life Survey will be used to compare QOL between Dapagliflozin vs Placebo.

OTHER OUTCOMES:
Effect of Dapagliflozin on change in Validated Echocardiographic Indices & Biomarkers of Atrial Myopathy | Baseline and 3 months
  To determine the effect of Dapagliflozin on validated echocardiographic indices and biomarkers of atrial myopathy in patients with AF and DM. We will compare left atrial volume index (ml/m2), left atrial strain and atrial tissue dopplers (cm/s). All measurements will be performed at baseline and at study completion and compared between Dapagliflozin vs Placebo. We will measure brain natriuretic peptide and other biomarkers as well.

CONTACTS AND LOCATIONS:
Overall Officials: Zain Ul Abideen Asad, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States